CLINICAL TRIAL: NCT02367495
Title: Trial of a Novel Paclitaxel-coated Balloon With Citrate Excipient for Restenosis in -Limus Analogue Drug-eluting Coronary Stents
Brief Title: Trial of a Novel Paclitaxel-coated Balloon With Citrate Excipient for Restenosis in -Limus Analogue DES
Acronym: ISAR-DESIRE 3A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No.S03814
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Coronary Restenosis
Keywords: Coronary Restenosis; restenosis; paclitaxel-coated balloon; drug-eluting stent; drug-coated balloon; coronary angiography
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCB (Experimental): Paclitacel-coated balloon (Agent, Boston Scientific)
  Interventions: Device: PCB

INTERVENTIONS:
Device: PCB — PCB with Citrate-based excipient

SUMMARY:
Hypothesis:

Angioplasty with a novel paclitaxel-coated balloon (PCB; Agent, Boston Scientific) with citrate-based excipient will be non-inferior to conventional paclitaxel-coated balloon with iopromide excipient (PCB) for the treatment of coronary restenosis after implantation of limus-analogue drug-eluting stents (DES)

DETAILED DESCRIPTION:
The optimal management of patients presenting with drug-eluting stent (DES) restenosis remains unclear. Data from recent randomized clinical trials have suggested that angioplasty with drug-coated balloons (DCB) is associated with excellent clinical outcomes. However, as the effectiveness of DCB devices depends critically on the specific composition of its matrix coating there may be important differences in clinical performance between different DCB devices. The prospective, non-randomized, single arm, historical-control ISAR-DESIRE 3A trial is designed to test that hypothesis that angioplasty with a novel paclitaxel-coated balloon with citrate-based excipient (Agent PCB, Boston Scientific) will be non-inferior to a conventional paclitaxel-coated balloon with iopromide excipient (SeQuent Please PCB, B. Braun; data from ISAR-DESIRE 3) for the treatment of coronary restenosis after implantation of limus-analogue drug-eluting stents (DES). The key inclusion criteria are patients with symptoms and/or objective signs of ischemia, restenosis at the site of previous limus-analogue DES implantation and written, informed consent. The primary endpoint is in-segment percent diameter stenosis (%DS) at 6-8 month follow-up angiography. Sample size calculation is based on a non-inferiority analysis: %DS of 35% after Both PCB, non-inferiority margin of 7% absolute, 1-sided α-level of 0.05 and power of 80% resulting in 102 patients per group. To account for possible FU losses 125 patients in total will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% restenosis after prior implantation of LES in native coronary vessels.
2. Written, informed consent by the patient for participation in the study.
3. In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

1. Age < 18 years
2. Cardiogenic shock
3. Acute ST-elevation myocardial infarction within 48 hours from symptom onset.
4. Target lesion located in the left main trunk or bypass graft.
5. Target lesion located in small vessel (vessel size < 2.0 mm)
6. Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
7. Severe renal insufficiency (glomerular filtration rate ≤ 30 ml/min)
8. Contraindications to antiplatelet therapy, paclitaxel
9. Pregnancy (present, suspected or planned) or positive pregnancy test.
10. Previous enrollment in this trial.
11. Patient's inability to fully comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
In-segment percent diameter stenosis (%DS) | at 6-8 months

SECONDARY OUTCOMES:
In-segment minimal lumen diameter and binary restenosis | at 6-8 months
Composite of death or myocardial infarction | at 12 months
Target lesion revascularization and thrombosis | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Byrne, MB BCh PhD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Koch T, Lenz T, Rheude T, Cassese S, Xhepa E, Joner M, Mehilli J, Schunkert H, Kastrati A, Kufner S. Comparative long-term efficacy and safety of two paclitaxel-coated balloons with different coating strategies for the treatment of drug-eluting coronary stent restenosis. Catheter Cardiovasc Interv. 2024 Nov;104(5):909-917. doi: 10.1002/ccd.31228. Epub 2024 Sep 18. PMID 39290129
- [Derived] Kufner S, Rai H, Wiebe J, Altevogt F, Pyxaras S, Joner M, Xhepa E, Cassese S, Colleran R, Schunkert H, Zrenner B, Kastrati A, Byrne RA; Intracoronary Stenting and Angiographic Results: Optimizing Treatment of Drug Eluting Stent In-Stent Restenosis 3A (ISAR-DESIRE 3A) Investigators. A prospective trial of a novel low-dose paclitaxel-coated balloon therapy in patients with restenosis in drug-eluting coronary stents Intracoronary Stenting and Angiographic Results: Optimizing Treatment of Drug Eluting Stent In-stent REstenosis 3A (ISAR-DESIRE 3A). Catheter Cardiovasc Interv. 2022 Feb;99(3):754-762. doi: 10.1002/ccd.30014. Epub 2021 Nov 18. PMID 34791755